CLINICAL TRIAL: NCT04305223
Title: Comparison of Dry Needling Versus Upper Extremity Strengthening and Dry Needling for Individuals With Cervicogenic Headache
Brief Title: Dry Needling for Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kathleen Geist, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00114985
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Headache; Cervicogenic Headache
Keywords: Headache; Dry Needling
MeSH Terms: conditions — Headache; Post-Traumatic Headache | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: single-blinded randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Investigators assessing outcome measures will be blinded to participants' group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling and upper extremity stretching program Arm (Experimental): Participants will receive a combination of dry needling and upper extremity stretching.
  * Dry needling in regions of the head and cervical spine will be positioned supine, sidelying or prone with the relevant myofascial trigger points treated using a Seirin L- type 30 mm needle (Seirin America, Inc., Weymouth, MA). The needle will be inserted to a depth no greater than three-quarters length of the needle for 30 seconds using a vertical pistoning technique and then statically up to 5 minutes.
  * A standard home exercise program consisting of strengthening and stretching exercises for the upper quarter.
  Interventions: Procedure: Dry Needling; Other: Upper extremity stretching program
- Dry Needling Arm (Active Comparator): Dry needling in regions of the head and cervical spine will be positioned supine, sidelying or prone with the relevant myofascial trigger points treated using a Seirin L- type 30 mm needle (Seirin American, Inc., Weymouth, MA). The needle will be inserted to a depth no greater than three-quarters length of the needle for 30 seconds using a vertical pistoning technique and then statically up to 5 minutes.
  Interventions: Procedure: Dry Needling

INTERVENTIONS:
Procedure: Dry Needling — Dry Needling is a treatment technique whereby a sterile, single-use, fine filament needle is inserted into the muscle to assist with decreasing pain and improving function through the release of myofascial trigger points (knots in the muscle).
  Other Names: Myofascial trigger point dry needling; Intramuscular stimulation
Other: Upper extremity stretching program — A standard home exercise program consisting of strengthening and stretching exercises for the upper quarter
  Arms: Dry needling and upper extremity stretching program Arm

SUMMARY:
This is a single-blinded randomized clinical trial. The primary aim of this study is to compare the effectiveness of dry needling of myofascial trigger points in the muscles of the head and cervical spine in addition to an upper extremity strengthening/stretching exercise program compared to a dry needling group alone on pain scores, cervical range of motion, pain sensitivity and changes in severity and frequency of pain symptoms in individuals with cervicogenic headache.

DETAILED DESCRIPTION:
This is a single-blinded randomized clinical trial. Eligible participants who agree to enroll in the study will be asked to attend four testing sessions. Participants in both groups will receive dry needling to the involved head and cervical muscles and the other group, in addition to receiving a dry needling intervention, will be instructed in a standard home exercise program consisting of strengthening and stretching exercises for the upper quarter. All dry needling (using standard clean technique) will be performed by licensed physical therapists board certified in orthopaedic physical therapy and having a minimum of 5 years of experience treating patient populations with dry needling.

The aim of this research study is to compare he effectiveness of dry needling alone with dry needling and a home exercise program on pain, pain sensitivity, cervical range of motion, and changes in the severity and frequency among individuals with headache symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral headache (HA) without side shift
* H/o pain triggered by neck movement
* Limitation in cervical range of motion
* Ispilateral neck, shoulder or arm pain
* Intermittent pain with episodes varying in duration
* Head and neck pain is non-throbbing in nature

Exclusion Criteria:

* Use of anti-coagulation medicine (except low dose aspirin)
* Pregnancy
* Acute or uncontrolled medical illness
* Opioid use within six months
* Fibromyalgia or diffuse painful syndromes in the UE or LE
* Substance abuse
* Presence of fever, vomiting or visual changes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Change in visual analog score for pain level | Baseline, Weeks 1 to 4 post intervention
  Pain is reported using a Visual Analog Scale from 0-10 and evaluates the frequency, severity and duration of the pain. Higher score indicates worse outcome.
Change in pain pressure threshold (PPT) | Baseline, Weeks 1 to 4 post intervention
  Pressure algometry is a method described to determine pressure pain threshold (PPT) by applying controlled pressure to a given body point. Measured with a pressure algometer: 0-50 KPa/s (kilopascal/second squared), minimum score representing increased pain to light touch/measuring allodynia.
Change in cervical range of motion | Baseline, Weeks 1 to 4 post intervention
  Will measure C1-2 Active Range of Motion, min score, 0; max score 50 degrees, lower score more limited (worse outcome).
Functional outcome measure: Change in neck disability index | Baseline, Weeks 1 to 4 post intervention
  Score ranges from 0-50 points: higher scores indicate higher levels of disability; Minimal detectable change (MDC), 5 points.
Functional outcome measure: Change in headache disability index | Baseline, Weeks 1 to 4 post intervention
  Score ranges from 0-72: 0 is no disability, 72 is more severe disability. Minimally Clinically Important Difference (MCID) is 29 points.
Change in Pain Frequency-Severity-Duration (PFDS) Scale | Baseline, Weeks 1 to 4 post intervention
  PFSD scale ranges from 1-140 with higher scores indicative of higher disability.
  There is a composite score that ranges from 0-140. Higher score correlates with worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Geist, PT, DPT, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States